CLINICAL TRIAL: NCT03984305
Title: Utilization of Target Ranges to Treat Patients With Parkinson's Disease by Objective Measurement Using the Personal KinetiGraph® (PKG®) Compared to Standard of Care Assessment (TARGET-PD)- A Randomized Controlled Trial
Brief Title: Utilization of Target Ranges to Treat Parkinson's Disease With the PKG
Acronym: TARGET-PD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to significant protocol updates that resulted in initiating a new study
Sponsor: Global Kinetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Study 003
Record Dates: First submitted 2019-06-07; First posted 2019-06-13 (Actual); Results first posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
Keywords: Personal KinetiGraph (PKG) Movement Recording System; Objective Measurement
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized using the Electronic Data Capture (EDC) system in a 1:1 ratio to the PKG- Group (standard of care clinical assessments without use of PKG data) or the PKG+ Group (standard of care clinical assessments plus use of PKG data).
Who Masked: Participant
Masking Description: Subjects will remain blinded to treatment group throughout the life of the trial. Investigator and research staff will be unblinded to the treatment group as they will or will not have access to the PKG results to be incorporated into their standard of care practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PKG+ Group (Experimental): For subjects in the PKG+ Group, participants will wear the PKG watch prior to all study visits in which the study investigator will review and report on the PKG prior to the visit and use the information to guide the discussion with the subject during the clinical assessment.The PKG will be used to determine if the subject is "controlled" or "uncontrolled" based on scores provided by the PKG.
  Interventions: Device: Personal KinetiGraph® (PKG®) Watch; Device: Personal KinetiGraph® (PKG®) Report
- PKG- Group (Placebo Comparator): For subjects in the PKG- Group (SOC control group), participants will wear the PKG watch prior to all study visits, however the investigator will not have access to the PKG report and will use standard of care to determine clinical treatment plans.
  Interventions: Device: Personal KinetiGraph® (PKG®) Watch

INTERVENTIONS:
Device: Personal KinetiGraph® (PKG®) Watch — The Personal KinetiGraph (PKG®) Movement Recording System consists of the following:
  * A wrist-worn data logger (PKG Watch) designed to acquire data on the kinematics of movement disorder symptoms over a 6-10 day period.
  * An application to configure the data logger and transfer the acquired data at the end of a recording.
Device: Personal KinetiGraph® (PKG®) Report — The Personal KinetiGraph (PKG®) Movement Recording System was developed by neurologists at the Melbourne-based Florey Institute of Neuroscience and Mental Health. The product is manufactured and marketed by GKC.
  The Personal KinetiGraph (PKG®) Movement Recording System consists of the following:
  • A series of algorithms that analyze the uploaded data, producing a PDF that is delivered to the clinician. The PDF contains objective data distinguishing the movement patterns consistent with tremor, bradykinesia, dyskinesia and immobility.
  Arms: PKG+ Group

SUMMARY:
The main objective of this study is to evaluate whether people whose PD symptoms are uncontrolled who are managed with the aid of objective measurement and use of target ranges have improved PD symptoms and outcomes as compared to individuals treated using only standard of care (medical history, neurological examination).

DETAILED DESCRIPTION:
This is a randomized controlled trial (RCT) to evaluate treating uncontrolled patients with Parkinson's Disease (PwP) to a target range as suggested by expert review papers. The study aims to evaluate clinical patient outcomes, quality of life measures and health care utilization of those patients specifically treated to a target range when using the PKG data in the clinical management of Parkinson's disease (PD) in routine clinical care (treatment group) compared to those managed with medical history and clinical evaluation alone (control group) performed by a neurologist experienced in PD management. Both groups will be recommended to undergo medication changes until they reach a "controlled state" that is determined by either the clinician using standard of care (SOC) (PKG- Group) or using PKG based targets and SOC assessments (PKG+ Group).

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign a written informed consent for study participation
* Presumed to have Levodopa responsive idiopathic Parkinson's Disease
* Age inclusive at the time of consent per PKG Indications for Use (46-83 years old)
* Has not been previously managed with the PKG

Exclusion Criteria:

* Contraindication to increasing levodopa (e.g. orthostatic hypotension, hallucinations/psychosis or any other medical condition in the last year that would preclude increasing levodopa or other appropriate Parkinson's Disease medications)
* MoCA score <23 at screening visit
* Diagnosis of Essential Tremor
* Wheelchair bound or bedridden
* Currently utilizing or planning in the next 6 months advanced PD therapies (DBS, infusion, etc.)
* In the investigator's or sponsor's opinion, subject has any unstable or clinically significant condition that would impair the participant's ability to comply with study requirements or interfere with interpretation of the study endpoints (e.g., subject unable to complete PKG watch wear instructions per Patient Instruction Manual)

Ages: 46 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raja Mehanna, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (17):
- United States (17):
  - Washington Regional Medical Center, Fayetteville, Arkansas
  - University of Arkansas Medical Center, Little Rock, Arkansas
  - Parkinson's Disease and Movement Disorders Center of Silicon Valley, Menlo Park, California
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kaiser Mid-Atlantic Permanente Center, Rockville, Maryland
  - Neurology Center of New England, Foxborough, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - University of Nebraska, Omaha, Nebraska
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Parkinson's Disease and Movement Disorders Center of Long Island, Commack, New York
  - Weill Cornell, New York, New York
  - University of Texas, Houston, Texas
  - Marshall University, Huntington, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pahwa R, Isaacson SH, Torres-Russotto D, Nahab FB, Lynch PM, Kotschet KE. Role of the Personal KinetiGraph in the routine clinical assessment of Parkinson's disease: recommendations from an expert panel. Expert Rev Neurother. 2018 Aug;18(8):669-680. doi: 10.1080/14737175.2018.1503948. Epub 2018 Jul 26. PMID 30032695
- [Background] Shulman LM, Gruber-Baldini AL, Anderson KE, Fishman PS, Reich SG, Weiner WJ. The clinically important difference on the unified Parkinson's disease rating scale. Arch Neurol. 2010 Jan;67(1):64-70. doi: 10.1001/archneurol.2009.295. PMID 20065131
- See also: Sponsor website — https://www.globalkineticscorporation.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- PKG+ Group: For subjects in the PKG+ Group, participants will wear the PKG watch prior to all study visits in which the study investigator will review and report on the PKG prior to the visit and use the information to guide the discussion with the subject during the clinical assessment.The PKG will be used to determine if the subject is "controlled" or "uncontrolled" based on scores provided by the PKG.
  Personal KinetiGraph® (PKG®) Watch: The Personal KinetiGraph (PKG®) Movement Recording System consists of the following:
  * A wrist-worn data logger (PKG Watch) designed to acquire data on the kinematics of movement disorder symptoms over a 6-10 day period.
  * An application to configure the data logger and transfer the acquired data at the end of a recording.
  Personal KinetiGraph® (PKG®) Report: The Personal KinetiGraph (PKG®) Movement Recording System was developed by neurologists at the Melbourne-based Florey Institute of Neuroscience and Mental Health. The product is manufactured and marketed by GKC.
  The Personal KinetiGraph (PKG®) Movement Recording System consists of the following:
  • A series of algorithms that analyze the uploaded data, producing a PDF that is delivered to the clinician. The PDF contains objective data distinguishing the movement patterns consistent with tremor, bradykinesia, dyskinesia and immobility.
- PKG- Group: For subjects in the PKG- Group (SOC control group), participants will wear the PKG watch prior to all study visits, however the investigator will not have access to the PKG report and will use standard of care to determine clinical treatment plans.
  Personal KinetiGraph® (PKG®) Watch: The Personal KinetiGraph (PKG®) Movement Recording System consists of the following:
  * A wrist-worn data logger (PKG Watch) designed to acquire data on the kinematics of movement disorder symptoms over a 6-10 day period.
  * An application to configure the data logger and transfer the acquired data at the end of a recording.
Period: Overall Study
Arm/Group | PKG+ Group | PKG- Group
Started | 23 | 18
Completed | 0 | 0
Not Completed | 23 | 18
Not completed — Sponsor Request due to Study Discontinuation | 19 | 15
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects enrolled prior to the early enrollment closure, and followed through the 4-month visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | PKG+ Group | PKG- Group | Total
Number analyzed (Participants) | 23 | 18 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.6 (4.4) | 71.4 (5.8) | 73.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 16 | 8 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 15 | 36
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 16 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 23 | 18 | 41
Years since Parkinson's Disease Diagnosis [Mean (Standard Deviation); unit: years] | 5.4 (4.7) | 6.3 (4.4) | 6.3 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Outcomes Using Movement Disorder Specialist - Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
Description: The change in total MDS-UPDRS score at 4 months from baseline defined as sections I, II, III and IV in Patients with Parkinson's. The endpoint will be compared between those who are treated with standard of care and access to the PKG (PKG+ Group) and those who are treated per standard of care alone (PKG- Group). The MDS-UPDRS evaluates motor and non-motor symptoms in persons with Parkinson's and consists of 4 parts with various questions and evaluations. Parts I and II (non-motor) each contain 13 questions/evaluations, Part III (motor) contains 33 and Part IV (motor) contains 6. Each question/evaluation score ranges from 0 (normal) to 4 (severe). Higher scores indicate a greater impact of Parkinson's disease symptoms (i.e., worse symptoms).
Time Frame: From Baseline to the 4 month Follow-up Visit (approximately 3-9 months)
Population: The primary analysis is based on the intent-to-treat population defined as all randomized subjects analyzed according to the treatment group assigned. Subjects were excluded from the analysis if they did not complete the 4 month Follow-up Visit or did not complete all parts of the MDS-UPDRS assessment at the Baseline and/or 4 month Follow-up Visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PKG+ Group | PKG- Group
Number analyzed (Participants) | 16 | 11
score on a scale | 0.9 (19.9) | 0.8 (12.0)

2. Secondary Outcome: Percentage of Responders for Total MDS-UPDRS
Description: Percent "responders" for total MDS-UPDRS based on a minimal clinically important change of 4.3 (Shulman LM, Gruber-Baldini AL, Anderson KE, et al. The Clinically Important Difference on the Unified Parkinson's Disease Rating Scale. Arch Neurol 2010: 67(1):64-70.)
Time Frame: 4 month Follow-up Visit
Population: The primary analysis is based on the intent-to-treat population defined as all randomized subjects analyzed according to the treatment group assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | PKG+ Group | PKG- Group
Number analyzed (Participants) | 16 | 11
Participants | 6 | 3

3. Secondary Outcome: Change in Parkinson's Disease Questionnaire-39 Questions (PDQ-39)
Description: Change in the patient reported quality of life questionnaire PDQ-39 from Baseline. The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality of life issues across 8 dimensions. Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better quality of life.
Time Frame: From Baseline to the 4 month Follow-up Visit (approximately 3-9 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PKG+ Group | PKG- Group
Number analyzed (Participants) | 19 | 15
score on a scale | 6.3 (17.5) | -1.5 (5.1)

4. Secondary Outcome: Change in MDS-UPDRS Total From Baseline
Description: as for outcome 1
Time Frame: From Baseline to the 1, 2 and 3-Year Annual Visits
Population: This Secondary Outcome Measure was not evaluated because the study was discontinued after completion of the 4-month Follow-up Visit. Subjects did not complete the 1, 2, or 3-Year Annual Follow-up Visits.
Arm/Group | PKG+ Group | PKG- Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in MDS-UPDRS Sub Part I
Description: Change in sub part I of the MDS-UPDRS from baseline. The MDS-UPDRS evaluates motor and non-motor symptoms in persons with Parkinson's and contains 4 sub parts. Each sub part is summed to give a total score MDS-UPDRS score. Sub part I assesses the non-motor impact of Parkinson's disease and contains 13 questions/evaluations. Each question/evaluation score ranges from 0 (normal) to 4 (severe). The minimum score for this sub part I is 0 and the maximum score is 52. Higher scores indicate a greater impact of Parkinson's disease symptoms (i.e., worse symptoms).
Time Frame: From Baseline to the 4 month Follow-up Visit (approximately 3-9 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PKG+ Group | PKG- Group
Number analyzed (Participants) | 18 | 15
score on a scale | -0.3 (4.7) | 1.1 (3.1)

6. Secondary Outcome: Change in PKG Bradykinesia Score (BKS)
Description: Change in the PKG reported scores BKS from baseline. Reported on a scale from 0-80. The higher the number, the more severe the bradykinesia.
Time Frame: From Baseline to the 4 month Follow-up Visit (approximately 3-9 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PKG+ Group | PKG- Group
Number analyzed (Participants) | 19 | 14
score on a scale | -1.4 (1.9) | -1.2 (2.5)

7. Secondary Outcome: Change in PKG Dyskinesia Score (DKS)
Description: Change in the PKG reported scores DKS from baseline. Reported on a scale of 0-355 with the higher the score, the more severe the dyskinesia.
Time Frame: From Baseline to the 4 month Follow-up Visit (approximately 3-9 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PKG+ Group | PKG- Group
Number analyzed (Participants) | 19 | 14
score on a scale | 0.1 (0.7) | 0.2 (1.3)

8. Secondary Outcome: Change in PKG Fluctuation Score (FDS)
Description: Change in the PKG reported scores FDS from baseline reported as a score of 0-45. The higher the score, the more severe the fluctuation.
Time Frame: From Baseline to the 4 month Follow-up Visit (approximately 3-9 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PKG+ Group | PKG- Group
Number analyzed (Participants) | 19 | 14
score on a scale | -0.2 (1.3) | -0.5 (1.6)

9. Secondary Outcome: Change in PKG Percent Time Tremor (PTT)
Description: Change in the PKG reported percent time in tremor from baseline, max 100%
Time Frame: From Baseline to the 4 month Follow-up Visit (approximately 3-9 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of time with tremor
Arm/Group | PKG+ Group | PKG- Group
Number analyzed (Participants) | 19 | 14
percentage of time with tremor | -1.6 (6.5) | -1.6 (5.9)

10. Secondary Outcome: Change in Levodopa Equivalent Dose (LED)
Description: Change in LED from baseline to 4-months
Time Frame: From Baseline to the 4 month Follow-up Visit (approximately 3-9 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: levodopa equivalent dose
Arm/Group | PKG+ Group | PKG- Group
Number analyzed (Participants) | 19 | 15
levodopa equivalent dose | 105.2 (229.5) | 61.7 (164.4)

11. Secondary Outcome: PKG Patient Survey
Description: Analyze PKG usability with the PKG Patient reported survey, specifically the percentage of subjects that strongly agree when asked if they would be willing to use the PKG again to assist in the management of Parkinson's disease. Questions in the survey are on a scale of strongly agree to strongly disagree and will be patient reported information related to their use of the PKG watch. Both treatment groups will be administered the survey and scores will be aggregated by group and compared.
Time Frame: Outcome measure evaluated at the 4-month Follow-up Visit
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PKG+ Group | PKG- Group
Number analyzed (Participants) | 19 | 15
Participants | 13 | 10

12. Secondary Outcome: Change in MDS-UPDRS Sub Part II
Description: Change in sub part II of the MDS-UPDRS from baseline. The MDS-UPDRS evaluates motor and non-motor symptoms in persons with Parkinson's and contains 4 sub parts. Each sub part is summed to give a total score MDS-UPDRS score. Sub part II assesses the non-motor impact of Parkinson's disease and contains 13 questions/evaluations. Each question/evaluation score ranges from 0 (normal) to 4 (severe). The minimum score for this sub part II is 0 and the maximum score is 52. Higher scores indicate a greater impact of Parkinson's disease symptoms (i.e., worse symptoms).
Time Frame: From Baseline to the 4 month Follow-up Visit (approximately 3-9 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PKG+ Group | PKG- Group
Number analyzed (Participants) | 18 | 15
score on a scale | 1.5 (7.2) | -1.3 (3.5)

13. Secondary Outcome: Change in MDS-UPDRS Sub Part III
Description: Change in sub part III of the MDS-UPDRS from baseline. The MDS-UPDRS evaluates motor and non-motor symptoms in persons with Parkinson's and contains 4 sub parts. Each sub part is summed to give a total score MDS-UPDRS score. Sub part III assesses the motor impact of Parkinson's disease and contains 33 questions/evaluations. Each question/evaluation score ranges from 0 (normal) to 4 (severe). The minimum score for this sub part III is 0 and the maximum score is 132. Higher scores indicate a greater impact of Parkinson's disease symptoms (i.e., worse symptoms).
Time Frame: From Baseline to the 4 month Follow-up Visit (approximately 3-9 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PKG+ Group | PKG- Group
Number analyzed (Participants) | 16 | 11
score on a scale | -1.6 (9.9) | -0.8 (8.3)

14. Secondary Outcome: Change in MDS-UPDRS Sub Part IV
Description: Change in Part IV of the MDS-UPDRS from Baseline. The MDS-UPDRS evaluates motor and non-motor symptoms in persons with Parkinson's and contains 4 sub parts. Each sub part is summed to give a total score MDS-UPDRS score. Sub part IV evaluates motor symptoms and contains 6 questions/evaluations. Each question/evaluation score ranges from 0 (normal) to 4 (severe). The minimum score for this sub part IV is 0 and the maximum score is 24. Higher scores indicate a greater impact of Parkinson's disease symptoms (i.e., worse symptoms).
Time Frame: From Baseline to the 4-month Follow-up Visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PKG+ Group | PKG- Group
Number analyzed (Participants) | 18 | 15
score on a scale | 0.1 (3.5) | 0.1 (2.0)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected at the time of enrollment through the 4-Month Follow-up Visits, which was a time period of approximately 1 year.
Description: Only the following protocol defined adverse events were collected during this post-market study: falls, orthostatic hypotension, bothersome hallucinations, delirium, impairment that prohibits interaction with the PKG Watch, hospitalizations, Emergency Department visits, urgent care visits and unanticipated clinic visits.
Arm/Group | PKG+ Group | PKG- Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/18
Serious Adverse Events (participants affected / at risk) | 3/23 | 1/18
Other Adverse Events (participants affected / at risk) | 12/23 | 3/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PKG+ Group (N=23) | PKG- Group (N=18)
Inpatient Hospitalization (Renal and urinary disorders) | 2 (2) | 1 (1) — Inpatient hospitalization due to either urinary tract infection(1), kidney stone(1) or ureteral mass with renal retention(1)
Inpatient Hospitalization (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PKG+ Group (N=23) | PKG- Group (N=18)
Fall (Injury, poisoning and procedural complications) | 6 (8) | 1 (1) — Fall that did not require medical attention or treatment
Orthostatic Hypotension (Vascular disorders) | 4 (6) | 2 (2) — Orthostatic Hypotension
Bothersome Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) — Bothersome Hallucinations
Emergency Room Visit (General disorders) | 1 (1) | 0 (0) — Emergency Room Visit due to neck pain
Urgent Care Visit (Infections and infestations) | 2 (2) | 0 (0) — Urgent Care Visit due to either sinusitis or upper respiratory infection
Unanticipated Clinic Visit (Gastrointestinal disorders) | 1 (1) | 0 (0) — Unanticipated Clinic Visit due to gastrointestinal pain

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A participating institution/PI may publish its individual site results; however, the sponsor has the exclusive right to publish the complete accumulated results of the multi-center trial. If a manuscript for the multi-center publication has not been submitted within 12 months of the conclusion or termination of the trial, then the institution/PI may publish a subset of the trial results. The sponsor shall be acknowledged in accordance with scientific practice.

DOCUMENTS (2):
  • Study Protocol (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT03984305/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT03984305/SAP_001.pdf